CLINICAL TRIAL: NCT02005159
Title: Study of the Impact of the Minimum Inhibitory Concentration and Susceptible Cut-off Points (CLSI, EUCAST and Pharmacokinetic/Pharmacodynamic) in Prognosis of Bacteremia by Enterobacteriaceae
Brief Title: Study of the Impact of the Minimum Inhibitory Concentration and Susceptible Cut-off Points (CLSI, EUCAST, and Pharmacokinetics/Pharmacodynamics)in Prognosis of Bacteremia by Enterobacteriaceae
Acronym: BACTERIEMIA
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-ANT-2011-01
Record Dates: First submitted 2013-11-14; First posted 2013-12-09 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Bacteremia by Enterobacteriaceae
Keywords: Enterobacteria; Bacteremia; Minimum inhibitory concentration; Susceptible; Prognosis
MeSH Terms: conditions — Bacteremia; Disease Susceptibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Positive blood-culture to bacteremia by enterobacteria: Patients with positive blood-culture to bacteremia by enterobacteria
  Interventions: Other: Microbiological studies

INTERVENTIONS:
Other: Microbiological studies

SUMMARY:
Provide scientific and validated data to help International Authorities to set susceptible to antibiotics cut-off points in bacteremia by Enterobacteriaceae

ELIGIBILITY:
Inclusion Criteria:

* >17 years old
* Clinically significant bacteremia
* Have received treatment fulfilling all this criteria:

  1. Treated with an only active antibiotic with enterobacteria (association with vancomycin, linezolid, daptomycin, metronidazole or clindamycin) between: cefotaxime, ceftriaxone, ceftazidime, cefepime, amoxicillin/clavulanic, piperacillin/tazobactam, ertapenem, imipenem, meropenem, ciprofloxacin or levofloxacin
  2. First antibiotic dose was administered during the first 12 hours after the time of sampling
  3. The antibiotic dosage was at least the advised amount in the summary of product characteristics to patient renal function
  4. The same antibiotic has been administered during at least 48 hours.

     Exclusion Criteria:

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bacteremia by Enterobacteriaceae attended in participants Hospitals during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correlation between the MIC of different antibiotics and the prognosis in patients with bacteremia. | 36 months
  Study the correlation between the minimum inhibitory concentration (MIC) of cefotaxime, ceftriaxone, cefepime, amoxicillin/clavulanic, piperacillin/tazobactam, ertapenem, imipenem, meropenem, ciprofloxacin and levofloxacin and the prognosis in patients with bacteremia by enterobacteria, with or without mechanisms of resistance
Correlation between CLSI and EUCAST cut-off points, FC/FD cut-off points with clinical prognosis and of the microbiological response in patients with bacteremia. | 36 months
  Determine if the CLSI and EUCAST (European Committee on Antimicrobial Susceptibility Testing) sensitive clinical cut-off points, as well as the suggested by pharmacokinetic and pharmacodynamic studies (FC/FD) are properly independent predictors of clinical prognosis and of the microbiological response in patients with bacteremia
Correlation between piperacillin/tazobactam serum concentrations and clinical prognosis | 36 months
  Evaluate if piperacillin/tazobactam serum concentrations are correlated with prognosis based on clinical sensitive cut-off points by CLSI and EUCAST

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez-Baño, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (14):
- Spain (14):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clínic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital San Pedro, Logroño
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- See also: Related Info — http://www.reipi.org/